CLINICAL TRIAL: NCT07375511
Title: The Contribution of Accelerated Recovery (mERAS) Approach to Postoperative Recovery in Pediatric Laparoscopic Surgery Cases
Acronym: Accelerated Re
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emel Yürük (Other)
Responsible Party: Sponsor-Investigator, Emel Yürük, ASSISTANT PROFESSOR, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ÇUKUROVA ÜNİVERSTY
Record Dates: First submitted 2025-12-24; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: mERAS Intervention; The ASA (American Society of Anesthesiologists) Score; The Patient Must be Between 4 and 12 Years Old
Keywords: Pediatric laparoscopic surgery; ERAS; Postoperative Recovery

STUDY DESIGN:
Intervention Model Description: This research was planned as a parallel-group, randomized controlled experimental study based on pre-test-post-test measurements to evaluate the effect of the Accelerated Recovery (mERAS) approach on postoperative pain, nausea-vomiting, thirst, fear, and recovery process in children undergoing pediatric laparoscopic surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mERAS Protocol Patient Group (Experimental): mERAS Protocol Patient Group
  Interventions: Other: mERAS Protocol
- Patient Group Receiving Standard Care (No Intervention): Preoperative Period: Within the scope of standard care, comprehensive education is not provided to patients and their families; only informed relatives are consulted to obtain surgical consent. During this period, patients' comorbidities are evaluated, and necessary medical treatments are applied. However, nutritional risk screening, which is emphasized in the literature, especially in pediatric surgery, is not routinely performed. While prophylactic antibiotic administration is aimed at, there is no standardized protocol for nausea-vomiting and pain management; treatment is carried out at the physician's discretion. Routine bowel preparation in accordance with current guidelines is not performed.

INTERVENTIONS:
Other: mERAS Protocol — mERAS Protocol Patient Group 1. Preoperative Period: Preparation and Education Within the scope of the mERAS protocol, both the child and their family are evaluated with a holistic approach in the preoperative period and prepared for the surgical process; this process is structured in accordance with the current ERAS guidelines for pediatric applications. Education and Counseling The child and their family will receive detailed information covering the preoperative, intraoperative, and postoperative processes. The child will be educated on preparing for the surgical experience using age-appropriate audiovisual materials; the family will be informed about the basic components of the recovery process, expected outcomes, and the contributions of the ERAS protocol. In addition, regular internal training for the surgeon, nurses, and anesthesia team will be provided to increase the applicability of the protocol and team cohesion. Preoperative Interventions
  • Patient and Family Information: P
  Arms: mERAS Protocol Patient Group

SUMMARY:
Pediatric laparoscopic surgery is a gold standard across all ages, offering benefits like smaller incisions, faster recovery, and better cosmetic outcomes. However, because children require more precise hemodynamic and respiratory management than adults, specialized perioperative care is essential. This study aims to evaluate the impact of a multidisciplinary Enhanced Recovery After Surgery (ERAS) approach on children aged 4-12, specifically measuring its effect on postoperative pain, nausea, thirst, fear levels, and the overall recovery process.

ELIGIBILITY:
Inclusion Criteria

* The patient must be between 4 and 12 years old,
* The ASA (American Society of Anesthesiologists) score must be 1 or 2,
* The parent(s) must be cognitively competent to give consent. Exclusion Criteria
* The child/parents must refuse to participate in the study,
* The presence of comorbidities that interfere with mobilization or oral feeding (which impairs the pain score),
* Chronic pain syndrome or regular opioid use,
* Previous major surgery in the same area (which may affect healing and pain experience).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale | 7 DAY
  Wong-Baker Faces Pain Rating Scale (Appendix 2): This is a visual self-assessment tool developed to evaluate the physical pain levels of individuals aged three years and older based on their own reports. The scale, consisting of six facial expressions, is scored from 0 = "no pain" to 10 = "very severe pain," and the child is asked to choose the face that best expresses the pain they are experiencing. It is a frequently used, valid, and understandable method for evaluating acute pain, especially in children who have difficulty verbally describing pain (Wong & Baker, 1988; Cohen et al., 2008).
  In this study, the postoperative pain levels of all children in the 4-12 age group will be evaluated using the Wong-Baker Faces Pain Rating Scale. In each measurement, the facial expressions will be explained to the children according to the standard instructions of the scale, and they will be asked to choose the face that best reflects the pain they are experiencing. The visual form of the scale
Baxter Animated Retching Faces Scale (BARF) | 7 days
  The Baxter Animated Retching Faces (BARF) Scale, developed by Baxter et al., is a self-report tool that assesses the severity of nausea using six-stage visual facial expressions ranging from "no nausea" to "severe nausea/vomiting." The faces on the scale are ordered to represent increasing levels of nausea (Baxter et al., 2011; Şişman et al., 2016).
Visual Thirst Scale | 7 days
  Visual Thirst Scale: The Visual Analog Scale (VAS) will be used to assess the severity of thirst in the postoperative period. On this scale, a value of 0 represents "no thirst" and a value of 10 represents "the most severe thirst the patient has ever felt." This approach is consistent with the method used by Conchon and Fonseca in their perioperative thirst studies to quantitatively assess the subjective severity of thirst (Conchon & Fonseca, 2015).
Children's Fear Scale | 7 days
  Children's Fear Scale: by McMurtry et al. (2011), the Children's Fear Scale is a visual self-assessment scale consisting of five facial expressions, scored between "no fear" (0) and "very frightened facial expression" (4), used to assess the level of fear experienced by children during medical procedures. The adaptation and validity-reliability study of the scale into Turkish was carried out by Gerçeker et al. (2018). No permission is required for clinical and research use of this scale (Children's Fear Scale - https://www.uoguelph.ca/pphc/childrens-fear-scale).

IPD SHARING:
Plan to Share IPD: No